CLINICAL TRIAL: NCT04631692
Title: Impact of Health Literacy Training for General Practitioners and a Consumer Facing Intervention to Improve Colorectal Cancer Screening in Underserved Areas: A Multicentric Cluster Randomized Controlled Trial
Brief Title: Evaluating a Health Literacy Intervention to Improve Colorectal Cancer Screening in Underserved Areas
Acronym: DECODE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Paul Sabatier of Toulouse (Other)
Collaborators: National Cancer Institute, France (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre Régional de Coordination des Dépistages des Cancers en Occitanie CRCDC-OC (Unknown); Aix Marseille Université (Other); Assistance Publique Hopitaux De Marseille (Other); Centre Régional de Coordination des Dépistages des Cancers Sud PACA (Unknown); Laboratoire HESPER-EA 7425 (Unknown); INSERM, UMR-S 1123 ECEVE Université de Paris (Unknown); Centre Régional de Coordination du dépistage des cancers - Ile-de-France (Unknown); University Paris 7 - Denis Diderot (Other); Centre Régional de Coordination du dépistage des cancers - Auvergne-Rhône-Alpes (Unknown); Institut Paoli-Calmettes (Other)
Responsible Party: Principal Investigator, Marie-Anne Durand, Researcher, University Paul Sabatier of Toulouse
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-A01687-32
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer Screening

STUDY DESIGN:
Intervention Model Description: We will use a two-arm randomized controlled cluster trial design trial with 8 clusters in total (2 clusters per region) and 4 general practitioners per cluster (i.e. 32 doctors in total). We will target disadvantaged areas in the following regions: Marseille, Lyon, Toulouse and Paris. We will use two ecological indexes of disadvantage: the European Deprivation Index (EDI) and the French Deprivation Index (FDEP). A community-based participatory research approach will be privileged throughout this project as well as focus groups and interviews
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking investigator, research assistants and data analyst
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (No Intervention): Usual care in participating primary care practices.
- Health literacy intervention (Active Comparator): Health literacy intervention combining health literacy and colorectal cancer screening training for general practitioners with a short brochure and video targeting eligible patients.
  Interventions: Behavioral: Health literacy intervention

INTERVENTIONS:
Behavioral: Health literacy intervention — We will translate and adapt an intervention developed by Ferreira et al. to address health literacy and improve CRC screening. This intervention combined a 2-hour health literacy training targeting primary care physicians (which also included information about CRC screening) and a patient level intervention that consisted of a brochure and video.
  In order to promote generalizability, large-scale diffusion, dissemination and sustained use beyond the funded-research period, we will use blended learning to develop a 2-hour e-learning health literacy training in French and a one-hour booster session.
  The patient-facing intervention (video + brochure) will follow key plain language and health literacy principles to translate evidence-based information in content that all patients can understand. Existing materials developed in France will be used and adapted as relevant.
  Arms: Health literacy intervention

SUMMARY:
The aim of this project is to assess the impact of a health literacy (HL) intervention combining HL and CRC screening training for general practitioners with a short brochure and video targeting eligible patients to increase CRC screening and other secondary outcomes in four underserved geographic areas in France. The investigators will use a two-arm randomized controlled cluster trial at 8 clusters (2 per area) primarily serving underserved populations across 4 geographic areas in France with 32 primary care physicians and 1024 patients recruited.

DETAILED DESCRIPTION:
Background Colorectal cancer (CRC) is a leading cause of cancer burden worldwide and the third most commonly diagnosed cancer in France (with 44,000 new cases in France each year). Systematic uptake of CRC screening can improve survival rates. However, people with limited health literacy (HL) and lower socioeconomic position rarely participate. The overall goal is to assess the impact of a HL intervention combining HL and CRC screening training for general practitioners with a short brochure and video targeting eligible patients to increase CRC screening and other secondary outcomes in four underserved geographic areas in France.

Methods The investigators will use a two-arm randomized controlled cluster trial at 8 clusters (2 per area) primarily serving underserved populations across 4 geographic areas in France with 32 primary care physicians and 1024 patients recruited. Primary care physicians practicing in underserved areas (identified using the European Deprivation Index and French Deprivation index) will be block-randomized to: 1) a combined intervention (HL and colorectal cancer training + brochure and video for eligible patients) or 2) usual care. The investigators will include all people between 50 and 74 years old who are eligible for CRC screening. The project will follow a community-based participatory research approach. The primary outcome is CRC screening uptake. The project will also include a qualitative needs assessment (focus groups and interviews) prior to finalizing the intervention and to test the acceptability of the combined intervention before the trial. After completing recruitment, semi-structured interviews will be conducted with up to 8 health professionals in each region (up to 24) and 6 to 12 patients per region (up to 48) based on data saturation. The investigators will explore strategies that promote the intervention's sustained use and rapid implementation using the Normalization Process Theory. A regression framework and mediation analyses will be used.

Discussion Limited HL and its impact on the general population is a growing public health and policy challenge worldwide. It has received limited attention in France. A combined HL intervention could reduce disparities in CRC screening, increase screening rates among most vulnerable populations, and increase knowledge and activation (beneficial in the context of repeat screening).

ELIGIBILITY:
Inclusion Criteria:

* People between 50 and 74 years old who are eligible for colorectal cancer screening and seen by a participating general practitioner.
* People who are able to complete a questionnaire in French, either alone or with help from a caregiver or relative.
* People with intellectual disability will be included as long as they are able to complete a questionnaire alone or with help from a caregiver or relative.

Exclusion Criteria:

- People whose mental health status does preclude participation in the study, as determined by the participating primary care practitioner or their qualified staff.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1025 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-12-07 (Actual); Study Completion 2025-04-14 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer screening uptake | up to 1-year post enrollment
  This information will be collected by each regional screening coordination center of the four participating regions, in collaboration with the health insurance (CPAM) at 6 months (for feedback to general practitioners in the intervention arm) and 1-year post enrollment into the study. It will also be collected using self-report in the patient questionnaire 1-year post enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Anne Durand, Principal Investigator — Université Toulouse III Paul Sabatier; Niamh M REDMOND, PhD, Principal Investigator — Université Toulouse III Paul Sabatier
Locations (4):
- France (4):
  - Service de recherche et épidémiologie cliniques, Lyon
  - Espace santé APHM, Marseille
  - Assistance Publique Hopitaux de Paris, Paris
  - Faculté de médecine, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Durand MA, Lamouroux A, Redmond NM, Rotily M, Bourmaud A, Schott AM, Auger-Aubin I, Frachon A, Exbrayat C, Balamou C, Gimenez L, Grosclaude P, Moumjid N, Haesebaert J, Massy HD, Bardes J, Touzani R, Diant LBEF, Casanova C, Seitz JF, Mancini J, Delpierre C. Impact of a health literacy intervention combining general practitioner training and a consumer facing intervention to improve colorectal cancer screening in underserved areas: protocol for a multicentric cluster randomized controlled trial. BMC Public Health. 2021 Sep 16;21(1):1684. doi: 10.1186/s12889-021-11565-3. PMID 34530800